CLINICAL TRIAL: NCT02991365
Title: Effekt Von Gewichtsabnahme Auf Die zentralnervöse Insulinresistenz Des Menschen
Brief Title: Effect of Weight Loss on Brain Insulin Sensitivity in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 8 weeks study
Record Dates: First submitted 2016-12-01; First posted 2016-12-13 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- nasal insulin (Active Comparator): daily administration of 160 U of human insulin as nasal spray
  Interventions: Other: nasal insulin
- placebo spray (Placebo Comparator): daily administration of placebo solution as nasal spray
  Interventions: Other: placebo spray

INTERVENTIONS:
Other: nasal insulin
  Arms: nasal insulin
Other: placebo spray
  Arms: placebo spray

SUMMARY:
Obesity if known to be associated with brain insulin resistance in humans. This condition has not only implication for the brain but also for whole-body energy homeostasis. Research in rodents indicates that weight loss is able to improve insulin sensitivity of the brain. The current project will test this hypothesis in humans. Therefore, brain insulin sensitivity will be assessed by fMRI in combination with intranasal insulin administration, using an established protocol. Furthermore, effects of daily administration of insulin nasal spray (versus placebo) over 8 weeks will be assessed as secondary (exploratory) variables.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c <6.5%
* Age between 40 and 75 years
* No intake of antidiabetic drugs or drugs for weight reduction
* no steroid intake
* Stable medication over 10 weeks before the start of the study

Exclusion Criteria:

* Persons who wear non-removable metal parts in or on the body.
* Persons with reduced temperature sensitivity and / or increased sensitivity to heating of the body
* Cardiovascular disease can not be ruled out, e.g. manifest coronary heart disease, heart failure greater than NYHA 2, previous heart attack, stroke condition
* Persons with hearing impairment or increased sensitivity to loud noises
* People with claustrophobia
* Minors or non-consenting subjects are also excluded
* Subjects with an operation less than 3 months
* Simultaneous participation in other studies
* Neurological and psychiatric disorders
* Subjects with hemoglobin Hb <11 g / dl
* Hypersensitivity to any of the substances used

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
brain insulin sensitivity | 30 minutes after administration of nasal insulin
  fMRI measurement will be performed before and after administration of 160 U of human insulin as nasal spray. Changes in regional activity will be quantified to assess regional brain insulin sensitivity.

SECONDARY OUTCOMES:
Effect of daily administration of 160 U nasal insulin or placebo over 8 weeks on body weight. | 8 weeks
  Participants will receive nasal insulin or placebo in a double-blind randomized fashion. Before and after 8 weeks body weight will be recorded.
Effect of daily administration of 160 U nasal insulin or placebo over 8 weeks on glucose tolerance . | 8 weeks
  Participants will receive nasal insulin or placebo in a double-blind randomized fashion. Before and after 8 weeks glucose tolerance will be assessed using a 75 g oral glucose tolerance test.
Effect of daily administration of 160 U nasal insulin or placebo over 8 weeks on body composition . | 8 weeks
  Participants will receive nasal insulin or placebo in a double-blind randomized fashion. Before and after 8 weeks body composition will be addressed by whole-body MRI and liver MRS.
whole-body insulin sensitivity | 2 hours
  Insulin sensitivity will be estimated from a frequent-sampling 75 g oral glucose tolerance test using the Matsuda formula.
Glucose tolerance | 2 hours
  a 75 g oral glucose tolerance test will be performed. Glucose tolerance will be defined by the American Diabetes Association criteria.
Cognitive function | 1 hours
  cognitive function will be addressed by neuropsychological testing.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fritsche, MD, Principal Investigator — University of Tübingen Hospital
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No